CLINICAL TRIAL: NCT02596529
Title: Medium-sized Posterior Fragments in AO-Weber B Fractures, Does Open Reduction and Internal Fixation Improve Outcome? A Multicenter Randomized Controlled Trial. The POSTFIX-trial.
Brief Title: Fixation of the Posterior Malleolus in Medium-sized Trimalleolar AO Weber-B Fractures.
Acronym: POSTFIX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Center Haaglanden (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Jochem Hoogendoorn, Dr., Medical Center Haaglanden
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL45763.098.13
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Trimalleolar Fracture; Posterior Malleolus; Open Reduction and Internal Fixation
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixation (Experimental): Patients with a medium-sized posterior fragment which will be treated by open reduction and internal fixation of all fractured malleoli.
  Interventions: Device: Fixation
- No fixation (Active Comparator): Patients with a medium-sized posterior fragment which will be treated bij open reduction and internal fixation of lateral and medial malleolus alone. No fixation of the posterior malleolus take place.
  Interventions: Other: NO Fixation

INTERVENTIONS:
Device: Fixation — Fixation of the posterior malleolus with lag-screws or platefixation (usually by Drittelrohr plate).
  Arms: Fixation
Other: NO Fixation — NO Fixation of the posterior malleolus.
  Arms: No fixation

SUMMARY:
The optimal treatment of ankle fractures with involvement of the posterior malleolus remains a subject of debate. Despite a large amount of literature on the role of the posterior malleolus in a so-called trimalleolar fracture, there are no clear guidelines for its treatment. Its size is the leading indication whether fixation of the fragment is necessary or not. Most orthopedic surgeons consider a posterior malleolar fracture fragment larger than 25% to 33% an indication for fixation. Interestingly, after careful evaluation of the available literature, there does not seem to be hard evidence for these numbers. It is generally accepted that restoration of a normal anatomic mortise and normal tibiotalar contact area are key elements for a good functional outcome. Inadequate reduction of the posterior fragment may alter the tibiotalar contact area and the joint biomechanics with altered stresses in parts of the joint, leading to the development of osteoarthritis and worse functional outcome. Traditionally, reduction of these larger fragments is indirectly, followed by percutaneous screw fixation in anterior-posterior direction. Disadvantages are that it is hard to achieve an anatomical reduction, and that fixation of smaller fragments is very difficult. Recently, a direct exposure of the posterior tibia via a posterolateral approach in prone position, followed by open reduction and fixation with screws in posterior-anterior direction or antiglide plate is advocated by several authors. This approach allows perfect visualization of the fracture, articular anatomical reduction, and strong fixation. Another advantage is that even small posterior fragments can be addressed. Several case series are published, which describe minimal major wound complications, good functional outcomes, and minimal need for reoperation. Since 2 years, in our institution we perform an open, anatomical reduction and fixation of all medium-sized posterior fragments via this approach. Although not thoroughly investigated yet, it seems to lead to better clinical outcomes than described in the literature and our retrospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* First ankle fracture of the affected side.
* Trimalleolar AO-Weber B fracture with additional medium-sized posterior fragment (5-25% of involved articular surface, AO type 44-B3)

Exclusion Criteria:

* severe traumatized patients
* Multiple fractures during visit emergency department
* Ankle fracture of the same ankle in the history
* Patients with pre-existent mobility problems
* Pre-existent disability
* Patients living in another region and follow-up will take place in another hospital.
* Inability to speak the dutch language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome 1 year after surgery measured by the AAOS-questionnaire (functional outcome of ankle/hindfoot in 27 questions) | 1 year

SECONDARY OUTCOMES:
Post-traumatic osteoarthritis 1 year after surgery measured by the Kellgren-Lawrence (1-4) score. | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - MCHaaglanden, The Hague, South Holland
  - Bronovo Ziekenhuis, The Hague, South Holland
  - Haga ziekenhuis, The Hague, South Holland

REFERENCES:
- [Derived] Verhage S, van der Zwaal P, Bronkhorst M, van der Meulen H, Kleinveld S, Meylaerts S, Rhemrev S, Krijnen P, Schipper I, Hoogendoorn J. Medium-sized posterior fragments in AO Weber-B fractures, does open reduction and fixation improve outcome? the POSTFIX-trial protocol, a multicenter randomized clinical trial. BMC Musculoskelet Disord. 2017 Feb 23;18(1):94. doi: 10.1186/s12891-017-1445-0. PMID 28231779